CLINICAL TRIAL: NCT04897334
Title: Transcranial Direct Current Stimulation and Rehabilitation to Ameliorate Impairments in Neurocognition After Stroke (TRAINS): Neuromodulatory Intervention to Ameliorate Cognition After Stroke for Individuals At Risk for VCID.
Brief Title: Transcranial Direct Current Stimulation and Rehabilitation to Ameliorate Impairments in Neurocognition After Stroke
Acronym: TRAINS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Kelly Sloane, MD, Assistant Professor of Neurology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 848469
Record Dates: First submitted 2021-05-17; First posted 2021-05-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke; Cognitive Impairment
Keywords: post-stroke cognitive impairment; transcranial direct current stimulation; neurorehabiliation
MeSH Terms: conditions — Ischemic Stroke; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcranial Direct Current Stimulation (tDCS) + cognitive therapy (Active Comparator): Participants will undergo 5 daily sessions of tDCS for 20 minutes using a montage in which an anode (2 mA) is placed over left dorsolateral prefrontal cortex and the cathode will be place on the right supraorbital area. Subjects will participate in cognitive therapy during stimulation.
  Interventions: Device: tDCS; Behavioral: Cognitive Therapy
- Sham Transcranial Direct Current Stimulation (tDCS) + cognitive therapy (Sham Comparator): Participants will undergo 5 daily sessions of sham tDCS for 20 minutes using a montage in which an anode (2 mA) is placed over left dorsolateral prefrontal cortex and the cathode will be place on the right supraorbital area. Subjects will participate in cognitive therapy during stimulation.
  Interventions: Device: sham tDCS; Behavioral: Cognitive Therapy

INTERVENTIONS:
Device: tDCS — tDCS is a type of non-invasive brain stimulation in which small electrical currents are applied to the scalp via 2 electrodes. During sham stimulation, the current, 2 mA, will be delivered for a short amount of time and then turn-off. To deliver the current, electrodes that are placed in saline soaked sponges. They will be attached to the left side of your head; they will be held in place with an elastic cap. For both real and sham stimulation the electrodes will be placed on the scalp. Most people cannot tell the difference between real and sham stimulation.
  Arms: Transcranial Direct Current Stimulation (tDCS) + cognitive therapy
Device: sham tDCS — tDCS is a type of non-invasive brain stimulation in which small electrical currents are applied to the scalp via 2 electrodes. During sham stimulation, the current, 2 mA, will be delivered for a short amount of time and then turn-off. To deliver the current, electrodes that are placed in saline soaked sponges. They will be attached to the left side of your head; they will be held in place with an elastic cap. For both real and sham stimulation the electrodes will be placed on the scalp. Most people cannot tell the difference between real and sham stimulation.
  Arms: Sham Transcranial Direct Current Stimulation (tDCS) + cognitive therapy
Behavioral: Cognitive Therapy — During both the treatment and the sham intervention, participants will undero cognitive therapy training by performing the NBack task. In this sequential letter memory exercise participants are presented with sequential stimuli in the form of a series of letters. For each new stimulus they are asked to indicate if the current stimulus matches the stimulus from 2 trials prior. This exercise stimulates cognitive demand in working memory, executive function and attention and is correlated with dorsolateral prefrontal cortex activity.

SUMMARY:
The purpose of this study is to determine whether a non-invasive brain stimulation technique, transcranial direct current stimulation (tDCS), combined with traditional cognitive therapy will improve cognitive function in patients with subacute stroke.

DETAILED DESCRIPTION:
This is a double-blind, sham-controlled study in which subjects with cognitive impairment after stroke will undergo neuropsychological testing before and after receiving 5 semi-consecutive daily sessions of real or sham transcranial direct current stimulation (tDCS) paired with cognitive therapy. Subjects will have experienced a stroke within 3 months of enrollment and will be undergoing inpatient rehabilitation at Penn Institute for Rehabilitation Medicine. Neuropsychological testing will be repeated immediately after completion of stimulation and 3-, 12- and 24- months following completion of treatment. The investigators will examine changes in cognitive performance induced by tDCS + cognitive therapy compared to sham tDCS + cognitive therapy. This study will combine knowledge gained from our behavioral, clinical and sociodemographic data in order to determine the relative degrees to which these properties predict whether persons with post-stroke cognitive impairment will respond to intervention.

ELIGIBILITY:
Inclusion Criteria:

* Stroke that occurred within 4 weeks of the study
* Presence of cognitive impairment attributable to stroke
* Between the ages of 18 and 90
* Able to understand the nature of the study and give informed consent
* Able to follow simple commands as evidenced by NIHSS subtest 1C =0

Exclusion Criteria

* History of chronic, serious, or unstable neurologic illness other than stroke
* Current unstable medical illness(es)
* History of reoccurring seizures or epilepsy
* Current abuse of alcohol or drugs (prescription or otherwise)
* Active and severe psychiatric disorder
* Metallic objects in the face or head other than dental apparatus such as braces, fillings, and implants.
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Baseline assessment prior to intervention; immediate post-intervention; 12 weeks (+/- 4 weeks) post-intervention; 12 months (+/- 4 weeks) post-intervention
  This psychometric test covers multiple domains of cognition, comes in multiple versions to avoid practice effect, is validated in the brain injury population and can be administered in 20-30 minutes. Possible scores on the RBANS range from 40 to 160 where a higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Sloane, MD, Principal Investigator — University of Pennsylvania; Roy Hamilton, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine Rehabilitation, Philadelphia, Pennsylvania, United States